CLINICAL TRIAL: NCT02181907
Title: Bioequivalence Study of UH-AC 62 XX Tablets 10 mg (TF4) Compared With the 10 mg Capsule Formulations Following Single Peroral Administration in Healthy Volunteers
Brief Title: Bioequivalence Study of UH-AC 62 XX Tablets Compared With the Capsule Formulations in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 107.260
Record Dates: First submitted 2014-07-02; First posted 2014-07-08 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-07

CONDITIONS: Healthy

ARMS (2):
- UH-AC 62 XX tablet (Experimental)
  Interventions: Drug: UH-AC 62 XX tablet; Drug: UH-AC 62 XX capsule
- UH-AC 62 XX capsule (Active Comparator)
  Interventions: Drug: UH-AC 62 XX tablet; Drug: UH-AC 62 XX capsule

INTERVENTIONS:
Drug: UH-AC 62 XX tablet
Drug: UH-AC 62 XX capsule

SUMMARY:
Study to investigate the bioequivalence of UH-AC 62 XX tablets 10 mg (TF4) and UH-AC 62 XX capsules 10 mg by single administration in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 20 and ≤ 35 years
* Weight : Body Mass Index ≥ 18.5 and < 25
* Subjects who are judged by the investigator to be appropriate as the subjects of the study based on results of screening test
* Subjects who volunteer to participate and are able to fully understand and agree to this study by written informed consent

Exclusion Criteria:

* History of gastrointestinal ulcer or surgery of gastrointestinal tract (except appendectomy)
* History of hypersensitivity to UH-AC 62 XX (meloxicam) or salicylate (aspirin etc.) or Non-steroidal anti-inflammatory drugs (NSAIDs)
* History of aspirin induced asthma (bronchial asthma induced by NSAIDs)
* A tendency of bleeding
* History of alcohol or drug abuse
* Taking an investigational drug within 4 months prior to the trial
* Whole blood donation more than 400 mL within 3 months prior to the trial
* Whole blood donation more than 100 mL within 1 month prior to the trial
* Donation of constituent of blood of more than 400 mL within 1 month prior to the trial
* Any medication which could influence the results of the trial within 10 days prior to the trial
* Excessive physical activities within 7 days prior to the trial
* Alcohol drinking within 3 days prior to the trial
* History of orthostatic hypotension, fainting spells or blackouts
* Other than above, those who were judged by the investigator to be inappropriate as the subjects of the study

Ages: 20 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2003-03; Primary Completion 2003-04 (Actual)

PRIMARY OUTCOMES:
Cmax (Maximum observed concentration of the analyte in plasma) | up to 60 hours after drug administration
AUC 0-60hr (Area under the concentration time curve of the analyte in plasma from zero time to 60 hours) | up to 60 hours after drug administration

SECONDARY OUTCOMES:
Tmax (Time to reach Cmax) | up to 60 hours after drug administration
t1/2 ( Terminal half-life of the analyte in plasma) | up to 60 hours after drug administration
AUC 0-infinity (Area under the concentration time curve of the analyte in plasma from zero time to infinity) | up to 60 hours after drug administration
MRTpo (Mean residence time of the analyte in the body after single dose po administration) | up to 60 hours after drug administration
Number of patients with adverse events | up to 20 days after final drug administration